CLINICAL TRIAL: NCT04073615
Title: Phase 1b/2 Open-label Study to Evaluate the Safety, Tolerability and Efficacy of Rivoceranib or Trifluridine/Tipiracil as Monotherapies and Rivoceranib and Trifluridine/Tipiracil as Combination Therapy in Subjects With Metastatic Colorectal Cancer
Brief Title: A Study of Rivoceranib and Trifluridine/Tipiracil for Metastatic Colorectal Cancer (mCRC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase 2 portion of the study was not performed due to redirection of the rivoceranib development plan by the Sponsor.
Sponsor: Elevar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RM-110
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rivoceranib (Experimental): Participants will receive an oral dose of rivoceranib once per day on Days 1 through 28 of each 28-day cycle.
  Interventions: Drug: Rivoceranib
- Trifluridine/tipiracil (Active Comparator): Participants will receive an oral dose of Trifluridine/tipiracil twice per day with food, on Days 1 through 5 and Days 8 through 12 of each 28-day cycle.
  Interventions: Drug: Trifluridine/Tipiracil
- Rivoceranib and trifluridine/tipiracil (Experimental): Participants will receive a daily oral dose of rivoceranib on Days 1 through 28 and the recommended phase 2 dose (RP2D) of trifluridine/tipiracil twice per day between Days 1 to 5 and 8 to 12 of each 28-day cycle.
  Interventions: Drug: Rivoceranib; Drug: Trifluridine/Tipiracil

INTERVENTIONS:
Drug: Rivoceranib — Film-coated tablets
  Other Names: Rivoceranib Mesylate; Apatinib Mesylate; Apatinib
  Arms: Rivoceranib; Rivoceranib and trifluridine/tipiracil
Drug: Trifluridine/Tipiracil — Film-coated tablets
  Other Names: Lonsurf
  Arms: Rivoceranib and trifluridine/tipiracil; Trifluridine/tipiracil

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose (RP2D) of rivoceranib when used in combination with trifluridine/tipiracil in participants with mCRC and to assess progression-free survival (PFS) in participants with mCRC.

DETAILED DESCRIPTION:
This a multicenter open-label study comparing safety, tolerability and efficacy of rivoceranib and trifluridine/tipiracil monotherapies, and the combination of rivoceranib plus trifluridine/tipiracil in participants with mCRC. Participants with histologically or cytologically definitive adenocarcinoma of the colon or rectum who have progressed following standard of care therapy for colorectal cancer (CRC) will be randomly assigned (1:1:2) to rivoceranib, trifluridine/tipiracil or rivoceranib plus trifluridine/tipiracil treatment groups.

The study will consist of an initial phase 1b portion to assess the safety of and determine the RP2D of rivoceranib in combination with trifluridine/tipiracil. A subsequent phase 2 portion will assess the primary endpoint of progression free survival (PFS) by investigator assessment. When a participant discontinues rivoceranib and/or trifluridine/tipiracil for any reason, the participant will enter the 12-month survival follow-up period until withdrawal of consent from the study, lost to follow-up, end of the study or death, whichever occurs earlier.

The maximum duration of the study is estimated to be 36 months, which includes screening, treatment, and follow-up phases.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of the diagnosis of mCRC
2. Failure to respond or be intolerant of at least 2 prior regimens of standard anti-cancer treatments (study treatment must be 3rd-line or greater for mCRC). Failed prior treatments may include:

   * Fluoropyrimidines-based chemotherapy
   * Irinotecan-based chemotherapy
   * Oxaliplatin-based chemotherapy
   * Anti-Vascular Endothelial Growth Factor (VEGF) biological therapy
   * Anti-Epidermal Growth Factor Receptor (EGFR) therapy, if RAS wild-type
   * Immunotherapy (for example, nivolumab, pembrolizumab and ipilimumab), in participants with Microsatellite Instability High/Deficient Mismatch Repair (MSI-H/dMMR). Participants who had received adjuvant chemotherapy and had recurrence during or within 6 months of completion of the adjuvant chemotherapy would be considered as 1 prior line of therapy
3. Have progressed based on imaging during or within 3 months of the last administration of most recent therapy
4. Have measurable disease, as defined by RECIST v1.1
5. Adequate bone marrow, renal, and hepatic function, as evidenced by the following within 7 days prior to Cycle 1 Day 1

   * Absolute neutrophil count (ANC) ≥1,500/mm3
   * Platelets ≥75,000/mm3
   * Hemoglobin ≥9.0 g/dL
   * Creatinine clearance (according to Cockcroft-Gault Equation or by 24 hr urine collection) > 50 mL/min and serum creatinine <1.0× upper limit of normal (ULN)
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3.0x ULN (≤5.0 × ULN for participants with liver involvement of their cancer)
   * Bilirubin ≤1.5 × ULN
   * Alkaline phosphatase ≤2.5 × ULN (≤5 × ULN with liver involvement of their cancer)
   * International normalized ratio (INR) / partial thromboplastin time (PTT) ≤1.5 × ULN (Participants currently under treatment with anti-thrombotic agents such as warfarin or heparin with no abnormal coagulation values can participate in this study)
6. Urinary protein <2+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates proteinuria ≥ 2+, a 24-hour urine or urine protein/creatinine ratio must be collected and must demonstrate <2 g of protein in 24 hours to allow participation in the study.
7. Have an Eastern Cooperative Oncology Group (ECOG) status of 0 or 1

Exclusion Criteria:

1. Prior treatment with rivoceranib or trifluridine/tipiracil
2. Prior treatment with other VEGFR small molecule inhibitors (for example, regorafenib)
3. Packed red blood cell transfusion or erythropoietin therapy within 14 days prior to first dose of study drug
4. History of another malignancy within 3 years prior to Cycle 1 Day 1. A participant with the following malignancies is eligible for this study if, in the opinion of the Investigator, they do not pose a significant risk to life expectancy:

   * Carcinoma of the skin without melanomatous features
   * Curatively treated cervical carcinoma in situ
   * Bladder tumors considered superficial such as noninvasive (T1a) and carcinoma in situ (Tis)
   * Thyroid papillary cancer with prior treatment
   * Prostate cancer which has been surgically or medically treated and not likely to recur within 3 years

6. Active renal dysfunction that requires dialysis treatments

7. Active cardiac disease including any of the following:

* Congestive heart failure New York Heart Association (NYHA) ≥Class 2
* Myocardial infarction less than 6 months before the start of Cycle 1 Day 1 of treatment

  8. Cardiac arrhythmias requiring antiarrhythmic therapy (beta-blockers or digoxin are permitted)

  9. History of uncontrolled hypertension (blood pressure ≥140/90 mmHg and/or change in antihypertensive medication within 7 days prior to first dose of study drug)

  10. History of antiangiogenic drug class-related severe adverse reactions, including uncontrolled hypertension or others related to prior therapy discontinuation and/or those that may indicate a higher risk to a participant' safety, in the Investigator's opinion, if provided further antiangiogenic treatment.

  11. History of vascular disease including arterial or venous embolic events (pulmonary embolism), other than hypertension, within 6 months prior to Cycle 1 Day 1 (for example, hypertensive crisis, hypertensive encephalopathy, stroke or transient ischemic attack [TIA], or significant peripheral vascular diseases) that, in the Investigator's opinion, may pose a risk to the participant on VEGF inhibitor therapy.

  12. History of clinically significant thrombosis within 3 months prior to first dose of study drug that, in the Investigator's opinion, may place the participant at risk of side effects from antiangiogenics medications

  13. History of bleeding diathesis or clinically significant bleeding within 14 days prior to first dose of study drug

  14. Therapy with systemic anticoagulant or antithrombotic agents within 7 days prior to first dose of study drug that in the Investigator's opinion could interfere with clotting. The maximum allowable daily dose of aspirin is 325 milligram (mg).

  15. Participants with unstable seizure disorder requiring medication changes within 3 months of Cycle 1 Day 1 treatment

  16. Untreated or active central nervous system (CNS) or leptomeningeal metastases. Participants are eligible if metastases have been treated and participants are neurologically returned to baseline or neurologically stable (expect for residual signs and symptoms related to the CNS treatment) for at least 4 weeks prior to first dose of study drug. In addition, participants must be either off corticosteroids, or on a stable dose or decreasing dose of ≤ 20 mg daily prednisone or prednisone-equivalent. A baseline radiological assessment of the brain will be performed on participants who have prior history of metastases with CNS involvement

  17. History of clinically significant glomerulonephritis, biopsy-proven nephritis, crystal nephropathy or other renal insufficiencies

  18. Unresolved adverse reactions >Grade 1 excluding peripheral neuropathy or treatment related myelosuppression

  19. Known hypersensitivity to any of the study drugs, study drug classes, or any components of study drug formulations

  20. Inability to swallow oral medications

  21. An active malabsorption condition, or any other condition that in the opinion of the Investigator might affect the absorption of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
(Phase 1b) Percentage of Participants with Dose-limiting Toxicity (DLT) During Cycle 1 | Baseline up to 28 days
(Phase 1b) Number of Participants with Adverse Events (AEs)investigator assessment | Baseline up to 3 years
(Phase 1b) Number of Participants with Serious Adverse Events (SAEs) | Baseline up to 3 years
(Phase 2) Progression Free Survival (PFS) per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by Investigator Assessment | Up to approximately 3 years

SECONDARY OUTCOMES:
(Phase 1b and Phase 2) Overall Survival (OS) | Up to approximately 3 years
  OS is the time from participant enrollment until death from any cause.
(Phase 2) Objective Response Rate (ORR) | Up to approximately 3 years
  ORR per RECIST v1.1 by Investigator Assessment is defined as percentage of participants who will achieve confirmed Complete Response (CR) or Partial Response (PR).
Duration of Response (DoR) | Up to approximately 3 years
  DoR per RECIST v1.1 by investigator assessment.
Time to Progression (TTP) | Up to approximately 3 years
  TTP per RECIST v1.1 by investigator assessment.
(Phase 2) Disease Control Rate (DCR) | Up to approximately 3 years
  DCR per RECIST v1.1 by investigator assessment.
(Phase 1b and 2) Number of Participants with Adverse Events (AEs) that Worsen in Severity as Defined by the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Florida Cancer Specialists, Sarasota, Florida
  - Northwestern University, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Vanderbilt University School of Medicine, Nashville, Tennessee